CLINICAL TRIAL: NCT03696342
Title: Clinical Study of the Efficacy of the Ophthalmic Solution of Pazufloxacin 0.6% (PRO-157) for the Treatment of Acute Bacterial Conjunctivitis, Compared to the Ophthalmic Solution of Gatifloxacin 0.3%.
Brief Title: Efficacy of the Ophthalmic Pazufloxacin 0.6% for Bacterial Conjunctivitis, Compared to Gatifloxacin 0.3%.
Acronym: PRO-157
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's convenience
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH157-0217/III
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-03

CONDITIONS: Conjunctivitis, Bacterial
Keywords: pazufloxacin; PRO-157; Fluoroquinolones
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — pazufloxacin; Gatifloxacin

STUDY DESIGN:
Intervention Model Description: clinical study of non-inferiority, multicenter, double-blind, with comparative group randomized
Who Masked: Participant, Investigator
Masking Description: In addition, the statistical analysis will be carried out in a blinded manner in the case of a partial and final analysis.
  The masking will be done using boxes in the primary packaging identical in the two groups and relabelling the bottles of both interventions.
  Blinding for the research subject and the researcher will be done by replacing the commercial labels in the case of the comparator in the bottles and the use of identical labels that contain the assignment number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-157 (Experimental): Pazufloxacin 0.6%. by Sophia Laboratories, topical ophthalmic
  1 drop, 3 times a day during the waking period in both eyes (at approximate intervals of 6 hours), for 7 days.
  Interventions: Drug: Pazufloxacin
- Zymar (Active Comparator): Gatifloxacin 0.3%. by Allergan, topical ophthalmic
  1 drop, 3 times a day during the waking period in both eyes (at approximate intervals of 6 hours), for 7 days.
  Interventions: Drug: Zymar

INTERVENTIONS:
Drug: Pazufloxacin — Pazufloxacin 0.6%. by Sophia Laboratories, topical ophthalmic
  1 drop, 3 times a day during the waking period in both eyes (at approximate intervals of 6 hours), for 7 days.
  Other Names: PRO-157
  Arms: PRO-157
Drug: Zymar — Gatifloxacin 0.3%. by Allergan, topical ophthalmic
  1 drop, 3 times a day during the waking period in both eyes (at approximate intervals of 6 hours), for 7 days.
  Other Names: gatifloxacin
  Arms: Zymar

SUMMARY:
Phase III clinical study of non-inferiority, multicenter, double-blind, with comparative group, of parallel groups and randomized. about a ophthalmic topical antibiotic for the treatment of bacterial conjunctivitis.

Goal:To compare the efficacy of the ophthalmic solution of pazufloxacin 0.6%, against the ophthalmic solution of gatifloxacin 0.3%, in the treatment of acute bacterial conjunctivitis.

Hypothesis:the ophthalmic solution PRO-157 is not inferior in the treatment of bacterial conjunctivitis, compared to the ophthalmic solution of gatifloxacin 0.3%, by means of the clinical remission of the disease.

Number of patients:

160 patients, each one will provide an eye for efficacy analysis, divided into 2 groups (80 eyes per group).

DETAILED DESCRIPTION:
The study subjects will be recruited from various research centers in western and central Mexico.

Each research center has a monitoring plan specified according to the recruitment capabilities of the same, which must be at least once a month, where the queries of your data entered into the electronic case report report will be reported to the center. (e-CRF) for which it has as time limit the next monitoring visit to make the pertinent changes.

The report of adverse events will be made according to the standard operating procedure (PNO) where it specifies, according to Official Mexican Standard 220 (NOM 220), that the signs or symptoms of adverse events will be reported based on the Medical Dictionary. for Regulatory Activities, for which the sponsor has version 20.1 in Spanish. For serious adverse events (SAEs) will be reported in accordance with the standardized operation procedure of pharmacovigilance of the sponsor, which adheres to the guidelines of NOM 220 and international regulations, these will be reported in the regulatory framework to the regulatory entity within a period of time no more than 7 days.

The study is registered in the National Registry of Clinical Trials (RNEC), entity equivalent to Clinical Trials in Mexico.

The quality assurance plan is carried out by the sponsor through the Quality Assurance agent in Clinical Research, whose function is to conduct inspections and audits of the research sites to document and generate reports of deviations from the protocol. In addition to the visits of the monitoring plan, the reliability of the data is guaranteed.

To verify the integrity, veracity and reliability of the data entered into the e-CRF, the monitors of each center will check the information uploaded to the portal with that reported in the source document of the principal investigator (PI), such as clinical notes, clinical history and documents. and formats attached to the research protocol, physical case report format, as well as those provided by the sponsor to the PI (subject's diary and quality and satisfaction survey).

The e-CRF used for this clinical study is provided by an internationally certified provider with the highest quality standards, protection of information under current regulations and confidentiality guarantee. The information that the PIs enter into the e-CRF is collated and verified by the clinical monitors and by the service provider's personnel, later reviewed and approved by the medical ophthalmologist researcher and by the Clinical Security Pharmacologist, who authorize the monitored data of clinical information and safety of the study molecule, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age ≥ 1 year.
* Both genders.
* Clinical picture of acute bacterial conjunctivitis defined by: Conjunctival secretion and conjunctival bulbar hyperemia

Exclusion Criteria:

* Pregnant women, lactating or planning to become pregnant.
* Women of reproductive age and who do not have a hormonal contraceptive method, intrauterine device or bilateral tubal obstruction.
* Participation in another clinical research study ≤ 30 days before the baseline visit.
* Previous participation in this same study.
* That they can not comply with their attendance at appointments or with all the requirements of the protocol.
* Single eye
* Presence of corneal abrasion or corneal ulceration in the study eye.
* History Users of contact lenses who are not willing to suspend their use during the study.
* Users of any formulation with ophthalmic application, including lubricants, that can not, or do not want to suspend it during the study.
* Antecedents of eye surgery 6 weeks prior to study entry.
* Viral or allergic conjunctivitis.
* Active uveitis.
* Active ulcerative keratitis.
* Recurrent corneal erosion syndrome
* Antecedent of hypersensitivity or allergy to fluoroquinolones.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (6):
- Mexico (6):
  - Consultorio Dra. Patricia Culebro Solano, Guadalajara, Jalisco
  - Juan Carlos Ochoa Tavares, Guadalajara, Jalisco
  - Samuel altamirano Vallejo, Guadalajara, Jalisco
  - Centro de investigación Medica Aguascalientes, Aguascalientes
  - Juan Carlos Serna Ojeda (INBIOMEDyC), Aguascalientes
  - Instituto Nacional de Pediatria, Mexico City

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- PRO-157: Pazufloxacin 0.6%. by Sophia Laboratories, topical ophthalmic 1 drop, 3 times a day during the waking period in both eyes (at approximate intervals of 6 hours), for 7 days.
  Pazufloxacin: Pazufloxacin 0.6%. by Sophia Laboratories, topical ophthalmic
  1 drop, 3 times a day during the waking period in both eyes (at approximate intervals of 6 hours), for 7 days.
- Zymar: Gatifloxacin 0.3%. by Allergan, topical ophthalmic 1 drop, 3 times a day during the waking period in both eyes (at approximate intervals of 6 hours), for 7 days.
  Zymar: Gatifloxacin 0.3%. by Allergan, topical ophthalmic
  1 drop, 3 times a day during the waking period in both eyes (at approximate intervals of 6 hours), for 7 days.
Period: Overall Study
Arm/Group | PRO-157 | Zymar
Started | 23; 23 Eyes | 23; 23 Eyes
Completed | 22; 22 Eyes | 23; 23 Eyes
Not Completed | 1; 1 Eyes | 0; 0 Eyes
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-157 | Zymar | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.78 (22.8) | 49.65 (29.2) | 48.22 (25.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 23 | 23 | 46
Concomitant medication [Count of Participants; unit: Participants] | 11 | 12 | 23
Positive culture [Count of Participants; unit: Participants] | 8 | 16 | 24
Severe conjunctival secretion [Count of Participants; unit: Participants] | 4 | 5 | 9
Severe bulbar conjunctival hyperemia [Count of Participants; unit: Participants] | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Amount of Conjunctival Secretion Present in Each Patient by the End of Treatment
Description: The ocular secretion will be classified as 0 = absent, 1 = mild, 2 = moderate and 3 = severe. The number will be reported according to the rating granted at final visit.
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-157 | Zymar
Number analyzed (Participants) | 22 | 23
Participants
  Absent | 20 | 21
  Mild | 2 | 2

2. Primary Outcome: Severeness of Conjunctival Bulbar Hyperemia in Each Patient by the End of Treatment
Description: Conjunctival hyperemia is defined as the simplest reaction of the conjunctiva to a stimulus, a red appearance secondary to the vasodilation of the conjunctival vessels of variable intensity. Will be graduated using the Efron scale.
  0 Normal , 1 Very slight, 2 Mild, 3 Moderate, 4 Severe.
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-157 | Zymar
Number analyzed (Participants) | 22 | 23
Participants
  Normal | 17 | 20
  Very mild | 5 | 3

3. Secondary Outcome: Overall Rating (Global Qualification) of Product's Efficacy as Classified by Main Investigator by the End of Treatment
Description: The global qualification of the investigator constitutes the integral judgment of the clinical picture of the subject, including signs and symptoms, after a routine ophthalmological evaluation and interrogation. It will be classified 0 = cure, 1 = improvement, 2 = no changes compared to before starting treatment, 3 = worsened. It will be registered in the CRF in each of the follow-up visits.
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-157 | Zymar
Number analyzed (Participants) | 22 | 23
Participants
  Cure | 16 | 19
  Improvement | 6 | 4

4. Secondary Outcome: Presence of Bacterial Eradication Compared to Baseline Culture Results
Description: The conjunctival secretion sample will be taken prior to the instillation of any medication, the result of the basal crop will be compared against the results of the final crop and the absence of bacterial species that were present in the culture of the baseline visit is considered bacterial eradication.
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-157 | Zymar
Number analyzed (Participants) | 22 | 23
Participants | 19 | 22

5. Secondary Outcome: Adverse Events
Description: The evaluation of adverse events requires a questioning conducted by the principal investigator and the appropriate exploratory techniques for its detection. the number of adverse events per study group will be considered for the analysis
Time Frame: day 0 to day 17 (visit 0 to security call)
Measure: Number; unit: number of adverse events
Arm/Group | PRO-157 | Zymar
Number analyzed (Participants) | 23 | 23
number of adverse events
  Mild Adverse Event | 25 | 27
  Moderate Adverse Event | 0 | 2

6. Secondary Outcome: Presence of Clinical Remission Defined as Absence of Hyperemia and Secretion by the Final Visit
Description: The clinical remission in the visits will be evaluated as "Yes" or "No", to report "Yes" it must have a grade of "0" in conjunctival hyperemia and "0" in secretion; otherwise, you must report as "No".
Time Frame: will be evaluated at the end of the treatment (day 8, final visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-157 | Zymar
Number analyzed (Participants) | 22 | 23
Participants | 15 | 19

ADVERSE EVENTS:
Time Frame: From day 1 (basal visit) to the safety call on day 15 (±2 days)
Description: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Arm/Group | PRO-157 | Zymar
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 20/23 | 18/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-157 (N=23) | Zymar (N=23)
Burning sensation (Eye disorders) | 19 (19) | 15 (15)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Ocular Pain (Eye disorders) | 0 (0) | 2 (2)
Blepharoedema (Eye disorders) | 0 (0) | 2 (2)
Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 1
Palpebral hyperemia (Eye disorders) | 0 (0) | 1 (1)
Ocular irritation (Eye disorders) | 0 (0) | 1 (1)
Tearing (Eye disorders) | 1 (1) | 1 (1)
Pruritus (Eye disorders) | 3 (3) | 3 (3)
Preexcitation syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Transparent Filament Presence (Eye disorders) | 1 (1) | 0 (0)
Ocular dryness (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial was terminated early due to the sponsor's convenience in the pipeline followed by the studied product. A small sample renders this results as merely descriptive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03696342/Prot_SAP_001.pdf